CLINICAL TRIAL: NCT04235673
Title: Oral Melatonin as Neuroprotectant in Preterm Infants .A Prospective, Double Blind vs Placebo, Parallel Arms Study
Brief Title: Oral Melatonin as Neuroprotectant in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesca Garofoli (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Sponsor-Investigator, Francesca Garofoli, PhD, Researcher, Co-PI,, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20180004210 17/01/2018
Record Dates: First submitted 2019-05-23; First posted 2020-01-22 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2022-10

CONDITIONS: Malondialdehyde; Melatonin
Keywords: Preterm neonate; Neuroprotection; Malondialdehyde; Melatonin
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melatonin (Experimental): melatonin oral drops; 3 mg/kg/day for 15 days
  Interventions: Dietary Supplement: melatonin
- placebo (Placebo Comparator): oral drops manufactured to mimic melatonin
  Interventions: Drug: placebo

INTERVENTIONS:
Dietary Supplement: melatonin — orally administered drops
  Other Names: not reported
  Arms: melatonin
Drug: placebo — orally administered drops
  Other Names: not reported
  Arms: placebo

SUMMARY:
Preterm newborns survival rates are improved, but long-term disabilities are still common. Major destructive focal lesions became less common, the most predominant lesion at present is diffuse white matter (WM damage). Melatonin (ME) serves as a neuroprotectant cerebral ischemia through its potent anti-oxidant/-inflammatory effect. Preclinical studies demonstrated that protects the developing brain by preventing abnormal myelination and inflammatory glial reaction. Clinical studies demonstrated ME ability in reducing brain damage after neonatal Hypoxic Ischemic Encephalopathy (HIE) or preventing neonatal impairments due to antenatal/ post-natal injuries: preeclampsia, IntraUterineGrowthRestriction (IUGR), ventilation, Bronchopulmonary Dysplasia (BPD). ME has a good safety profile with no known adverse effects. This study aims to highlight that ME can prevent brain impairment due to premature birth. ME will be administered orally (3 mg/kg/die for 15 days to neonates born before 29+6 week gestation, in a prospective double blind, randomized vs placebo study, 2 parallel arms. ME and malondialdehyde (MDA), a lipid peroxidation product) levels before and at the end of treatment will be measured . Other outcomes: Cerebral ultrasounds (cUS); cerebral magnetic resonance imaging (cMRI), " Fagan test " eye tracking, ophthalmological, auditory, neurological/cognitive child assessments. Monitoring parental distress, which can influence the neurodevelopmental outcome in preterms.

DETAILED DESCRIPTION:
About 552.000 infants are born in Italy each year, 1% of them with gestational age under 30 weeks. Survival rates are improved, but long-term disabilities are still common. Major destructive focal lesions became less common, the most predominant lesion at present is diffuse white matter (WM damage). The prevention of neurodevelopmental impairment is a major public health challenge and efforts are needed to test neuroprotective strategies. Melatonin (ME) serves as a neuroprotectant cerebral ischemia through its potent anti-oxidant/-inflammatory effect. Preclinical studies demonstrated that protects the developing brain by preventing abnormal myelination and inflammatory glial reaction. Clinical studies demonstrated ME ability in reducing brain damage after neonatal Hypoxic Ischemic Encephalopathy (HIE) or preventing neonatal impairments due to antenatal/ post-natal injuries: preeclampsia, IntraUterineGrowthRestriction (IUGR), ventilation, Bronchopulmonary Dysplasia (BPD). Ongoing studies are testing in premature neonates and pregnant women its neuroprotective properties. ME has a good safety profile with no known adverse effects.

This study aims to highlight that ME can prevent brain impairment due to premature birth. ME will be administered orally (3 mg/kg/die for 15 days within 96 hours from birth) to neonates born before 29+6 week gestation age (GA), in a prospective double blind, randomized vs placebo study, 2 parallel arms (30 preterm infants each). ME and malondialdehyde (MDA, a lipid peroxidation product) levels will be measured before and at the end of treatment. At birth, within 40 weeks of neonatal age, at 4-6 and at 24 months of age the following examinations are performed: Cerebral ultrasounds (cUS); cerebral magnetic resonance imaging (cMRI), during natural sleep (i.e. adopting sleep deprivation and/or feeding protocols); "Fagan test"eye tracking, ophthalmological, auditory brain stem evoked response (ABR), neurological/cognitive child assessments. Monitoring parental distress, which can influence the neurodevelopmental outcome in preterms.

ELIGIBILITY:
Inclusion Criteria

* preterm newborns gestational age GA < 29+6 weeks + day
* able to receive min 20ml/kg/day enteral nutrition, within 96 hours from birth
* written informed consent by both the parents.

Exclusion Criteria:

* preterm newborns GA > 29+6 weeks + days
* not able to receive enteral nutrition (min 20 ml/kg/die) within 96 hours of life
* infants with genetic and/or congenital metabolic or chronic diseases
* intraventricular hemorrhage (IVH) ≥ III,
* parents refusing to sign a written informed consent

Ages: 25 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde | 15 days
  plasmatic concentration pg/ml
Melatonin | 15 days
  plasmatic concentration pg/ml

SECONDARY OUTCOMES:
Cranial ultrasound (cUS) Assessment | up to 40 weeks
  to identify and score White Matter injuries
Brain Magnetic Resonance Immaging (cMRI) Assessment | up to 40 weeks
  Identify and score White Matter injuries
Auditory brain stem evoked response (ABR) Assessments | up to 40 weeks
  Identify and score auditory diseases

OTHER OUTCOMES:
Fagan Test of Infant Intelligence (FTII) | up to 24 months
  Measure the time ( minutes) to recognize unfamiliar versus familiar human faces to gauge visual-spatial encoding, attention, and working memory in infants.
Griffiths Mental Developmental Scales'Revised (GMDS-R) | up to 24 months
  The scales rate infant development across 5 main areas (locomotor, personal and social skills, hearing and language, eye and hand co-ordination, and performance), providing a general developmental quotient (DQ) of infants' abilities and 5 subscale quotients (SQ).
Child Behavior Checklist (CBCL) scales. | up to 24 months
  A self-rating scale to evaluate emotional, social, and behavioral problems in infants, according to the parents' evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Chryssoula Tzialla, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (4):
- Italy (4):
  - Child and Adolescence Neuropsychiatry Unit, Children's Hospital "Spedali Civili" of Brescia, 25123 Brescia, Italy., Brescia, BS
  - Neonatal Intensive Care Unit, Children's Hospital, University Hospital "Spedali Civili" Brescia, 25123 Brescia, Italy., Brescia, BS
  - Fondazione IRCCS Mondino, Pavia, PV
  - Neonatal Unit and NICU, Radiology, Clinical Chemistry Lab., Fondazione IRCCS Policlinico S. Matteo., Pavia, PV

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garofoli F, Longo S, Pisoni C, Accorsi P, Angelini M, Aversa S, Caporali C, Cociglio S, De Silvestri A, Fazzi E, Rizzo V, Tzialla C, Zecca M, Orcesi S. Oral melatonin as a new tool for neuroprotection in preterm newborns: study protocol for a randomized controlled trial. Trials. 2021 Jan 22;22(1):82. doi: 10.1186/s13063-021-05034-w. PMID 33482894